CLINICAL TRIAL: NCT02998528
Title: Randomized, OpenLabel, Phase 3 Trial of Nivolumab Plus Ipilimumab or Nivolumab Plus Platinum Doublet Chemotherapy Versus Platinum Doublet Chemotherapy in Early Stage NSCLC
Brief Title: A Neoadjuvant Study of Nivolumab Plus Ipilimumab or Nivolumab Plus Chemotherapy Versus Chemotherapy Alone in Early Stage Non-Small Cell Lung Cancer (NSCLC)
Acronym: CheckMate 816
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-816; 2016-003536-21 (EudraCT Number)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Cisplatin; Vinorelbine; Gemcitabine; Docetaxel; Pemetrexed; Carboplatin; Paclitaxel; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Platinum doublet chemotherapy (Active Comparator): Specified dose on specified days
  Interventions: Drug: Cisplatin; Drug: Vinorelbine; Drug: Gemcitabine; Drug: Docetaxel; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel
- Nivolumab plus platinum doublet chemotherapy (Experimental): Specified dose on specified days
  Interventions: Biological: Nivolumab; Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel
- Nivolumab plus Ipilimumab (Experimental): Specified dose on specified days
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Nivolumab plus Ipilimumab; Nivolumab plus platinum doublet chemotherapy
Drug: Cisplatin — Specified dose on specified days
  Arms: Nivolumab plus platinum doublet chemotherapy; Platinum doublet chemotherapy
Drug: Vinorelbine — Specified dose on specified days
  Arms: Platinum doublet chemotherapy
Drug: Gemcitabine — Specified dose on specified days
  Arms: Nivolumab plus platinum doublet chemotherapy; Platinum doublet chemotherapy
Drug: Docetaxel — Specified dose on specified days
  Arms: Platinum doublet chemotherapy
Drug: Pemetrexed — Specified dose on specified days
  Arms: Nivolumab plus platinum doublet chemotherapy; Platinum doublet chemotherapy
Drug: Carboplatin — Specified dose on specified days
  Arms: Nivolumab plus platinum doublet chemotherapy; Platinum doublet chemotherapy
Drug: Paclitaxel — Specified dose on specified days
  Arms: Nivolumab plus platinum doublet chemotherapy; Platinum doublet chemotherapy
Biological: Ipilimumab — This arm is closed and no longer enrolling patients.
  Other Names: BMS-734016; Yervoy
  Arms: Nivolumab plus Ipilimumab

SUMMARY:
The purpose of this neoadjuvant study is to compare nivolumab plus chemotherapy and chemotherapy alone in terms of safety and effectiveness, and to describe nivolumab plus ipilimumab's safety and effectiveness in treating resectable NSCLC.

This study has multiple primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Early stage IB-IIIA, operable non-small cell lung cancer, confirmed in tissue
* Lung function capacity capable of tolerating the proposed lung surgery
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Available tissue of primary lung tumor

Exclusion Criteria:

* Presence of locally advanced, inoperable or metastatic disease
* Participants with active, known or suspected autoimmune disease
* Prior treatment with any drug that targets T cell co-stimulations pathways (such as checkpoint inhibitors)

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2024-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (138):
- United States (57):
  - Local Institution - 0121, Glendale, Arizona
  - Local Institution - 0081, Los Angeles, California
  - Local Institution - 0025, Denver, Colorado
  - Local Institution - 0007, Plainville, Connecticut
  - Local Institution - 0173, Hollywood, Florida
  - Local Institution - 0136, Miami, Florida
  - Local Institution - 0054, Orlando, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Indian River Medical Center, Vero Beach, Florida
  - Northwest Georgia Oncology Center, P.C., Marietta, Georgia
  - Local Institution - 0015, Chicago, Illinois
  - Local Institution - 0002, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Local Institution - 0171, Fort Wayne, Indiana
  - Local Institution - 0170, Lexington, Kentucky
  - Local Institution - 0186, Louisville, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Local Institution - 0151, Baltimore, Maryland
  - Local Institution - 0001, Baltimore, Maryland
  - Local Institution - 0008, Boston, Massachusetts
  - Southcoast Center For Cancer, Fairhaven, Massachusetts
  - Local Institution - 0006, Newton, Massachusetts
  - Local Institution - 0012, Detroit, Michigan
  - Local Institution - 0090, Hattiesburg, Mississippi
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Local Institution - 0032, Las Vegas, Nevada
  - Local Institution - 0009, Hackensack, New Jersey
  - Valley Hospital Luckow Pavili, Westwood, New Jersey
  - Local Institution - 0027, Albany, New York
  - Local Institution - 0011, New York, New York
  - Local Institution - 0140, High Point, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Local Institution - 0149, Zanesville, Ohio
  - Kaiser Permanente, Portland, Oregon
  - Local Institution - 0139, Portland, Oregon
  - Local Institution - 0010, Philadelphia, Pennsylvania
  - Local Institution - 0018, Pittsburgh, Pennsylvania
  - Local Institution - 0013, Charleston, South Carolina
  - Local Institution - 0021, Charleston, South Carolina
  - Local Institution - 0146, Greenville, South Carolina
  - Local Institution - 0092, Nashville, Tennessee
  - Local Institution - 0005, Nashville, Tennessee
  - Local Institution - 0035, Austin, Texas
  - Texas Oncology, Bedford, Texas
  - Local Institution - 0153, Fort Bliss, Texas
  - Local Institution - 0106, Houston, Texas
  - Southwest Cancer Center, Lubbock, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Local Institution - 0143, Tyler, Texas
  - Local Institution - 0026, Waco, Texas
  - Intermountain Medical Center, Murray, Utah
  - Local Institution - 0003, Salt Lake City, Utah
  - Southwest Regional Cancer Clinic, St. George, Utah
  - Local Institution - 0135, Burlington, Vermont
  - Local Institution - 0125, Fairfax, Virginia
  - Local Institution - 0198, Fredericksburg, Virginia
- Argentina (2):
  - Local Institution - 0022, Capital Federal, Buenos Aires
  - Local Institution - 0023, Ciudad Autonoma de Buenos Aire, Buenos Aires
- Brazil (6):
  - Local Institution - 0079, Brasília, Federal District
  - Local Institution - 0077, Belo Horizonte, Minas Gerais
  - Local Institution - 0076, Ijuí, Rio Grande do Sul
  - Local Institution - 0073, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio Xii Hosp Cancer De Barretos, Barretos, São Paulo
  - Local Institution - 0075, Rio de Janeiro
- Canada (5):
  - Local Institution - 0095, Gatineau, Quebec
  - Local Institution - 0138, Montreal, Quebec
  - Local Institution - 0017, Montreal, Quebec
  - Local Institution - 0052, Trois-Rivières, Quebec
  - Local Institution - 0016, Saskatoon, Saskatchewan
- China (19):
  - Local Institution - 0161, Beijing, Beijing Municipality
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution - 0156, Beijing, Beijing Municipality
  - Local Institution - 0190, Guangzhou, Guangdong
  - Local Institution - 0192, Changsha, Hunan
  - Local Institution - 0175, Changsha, Hunan
  - Local Institution - 0193, Changsha, Hunan
  - Local Institution - 0179, Nanchang, Jiangxi
  - Local Institution - 0166, Nanchang, Jiangxi
  - Local Institution, Changchun, Jilin
  - Local Institution - 0159, Xi'an, Shan1xi
  - Local Institution - 0180, Xi'an, Shan3xi
  - Local Institution - 0160, Shanghai, Shanghai Municipality
  - Local Institution - 0178, Chengdu, Sichuan
  - Local Institution - 0163, Tianjin, Tianjin Municipality
  - Local Institution - 0189, Hangzhou, Zhejiang
  - Local Institution - 0183, Hangzhou, Zhejiang
  - Local Institution - 0182, Hangzhou, Zhejiang
  - Local Institution - 0165, Shanghai
- France (8):
  - Local Institution - 0059, Marseille
  - Local Institution - 0060, Paris
  - Local Institution - 0112, Paris
  - Local Institution - 0064, Pierre Benite Cedax
  - Local Institution - 0061, Rennes
  - Local Institution - 0113, Strasbourg
  - Local Institution - 0058, Toulouse
  - Local Institution - 0062, Tours
- Greece (2):
  - Local Institution - 0019, Athens
  - Local Institution - 0122, Thessaloniki
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Székesfehérvár
- Italy (5):
  - Local Institution - 0068, Bari
  - Local Institution - 0080, Genova
  - Local Institution - 0070, Perugia
  - Local Institution - 0066, Ravenna
  - Local Institution - 0067, Roma
- Japan (16):
  - Local Institution - 0131, Nagoya, Aichi-ken
  - Local Institution - 0118, Kashiwa-shi, Chiba
  - Local Institution - 0111, Kitakyushu-shi, Fukuoka
  - Local Institution - 0110, Fukushima, Fukushima
  - Local Institution - 0109, Hiroshima, Hiroshima
  - Local Institution - 0147, Sapporo, Hokkaido
  - Local Institution - 0133, Kobe, Hyōgo
  - Local Institution - 0123, Yokohama, Kanagawa
  - Local Institution - 0148, Sendai, Miyagi
  - Local Institution - 0127, Osaka, Osaka
  - Local Institution - 0119, Sakai-shi, Osaka
  - Local Institution - 0132, Sunto-gun, Shizuoka
  - Local Institution - 0126, Bunkyo-ku, Tokyo
  - Local Institution - 0120, Shinjuku-ku, Tokyo
  - Local Institution - 0108, Osaka
  - Local Institution - 0124, Tokyo
- Romania (3):
  - Local Institution - 0050, Craiova
  - Local Institution - 0051, Romania
  - Local Institution - 0069, Sector 2
- South Korea (3):
  - Local Institution - 0097, Busan
  - Local Institution - 0098, Hwasun
  - Local Institution - 0105, Seoul
- Spain (3):
  - Local Institution - 0028, Barcelona
  - Local Institution - 0029, Madrid
  - Local Institution - 0031, Majadahonda - Madrid
- Taiwan (4):
  - Local Institution - 0102, New Taipei City
  - Local Institution - 0107, Taichung
  - Local Institution - 0099, Taipei
  - Local Institution - 0100, Taipei
- Turkey (Türkiye) (3):
  - Local Institution - 0093, Adana
  - Local Institution - 0084, Ankara
  - Local Institution - 0115, Istanbul

REFERENCES:
- [Derived] Forde PM, Spicer JD, Provencio M, Mitsudomi T, Awad MM, Wang C, Lu S, Felip E, Swanson SJ, Brahmer JR, Kerr K, Taube JM, Ciuleanu TE, Tanaka F, Saylors GB, Chen KN, Ito H, Liberman M, Martin C, Broderick S, Wang L, Cai J, Duong Q, Meadows-Shropshire S, Fiore J, Bhatia S, Girard N; CheckMate 816 Investigators. Overall Survival with Neoadjuvant Nivolumab plus Chemotherapy in Lung Cancer. N Engl J Med. 2025 Aug 21;393(8):741-752. doi: 10.1056/NEJMoa2502931. Epub 2025 Jun 2. PMID 40454642
- [Derived] Awad MM, Forde PM, Girard N, Spicer J, Wang C, Lu S, Mitsudomi T, Felip E, Broderick SR, Swanson SJ, Brahmer J, Kerr K, Saylors GB, Chen KN, Gharpure V, Neely J, Balli D, Hu N, Provencio Pulla M. Neoadjuvant Nivolumab Plus Ipilimumab Versus Chemotherapy in Resectable Lung Cancer. J Clin Oncol. 2025 Apr 20;43(12):1453-1462. doi: 10.1200/JCO-24-02239. Epub 2025 Jan 8. PMID 39778121
- [Derived] Deutsch JS, Cimino-Mathews A, Thompson E, Provencio M, Forde PM, Spicer J, Girard N, Wang D, Anders RA, Gabrielson E, Illei P, Jedrych J, Danilova L, Sunshine J, Kerr KM, Tran M, Bushong J, Cai J, Devas V, Neely J, Balli D, Cottrell TR, Baras AS, Taube JM. Association between pathologic response and survival after neoadjuvant therapy in lung cancer. Nat Med. 2024 Jan;30(1):218-228. doi: 10.1038/s41591-023-02660-6. Epub 2023 Oct 30. PMID 37903504
- [Derived] Akinboro O, Drezner N, Amatya A, Runyan J, Fourie-Zirkelbach J, Zhao M, Bi Y, Korsah K, Mixter B, Tang S, Larkins E, Pazdur R, Beaver JA, Singh H. US Food and Drug Administration Approval Summary: Nivolumab Plus Platinum-Doublet Chemotherapy for the Neoadjuvant Treatment of Patients With Resectable Non-Small-Cell Lung Cancer. J Clin Oncol. 2023 Jun 10;41(17):3249-3259. doi: 10.1200/JCO.22.02509. Epub 2023 May 4. PMID 37141544
- [Derived] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N. Plain language summary of the CheckMate 816 study results: nivolumab plus chemotherapy given before surgery for non-small-cell lung cancer. Future Oncol. 2023 Mar;19(8):549-557. doi: 10.2217/fon-2023-0007. Epub 2023 Feb 23. PMID 36815433
- [Derived] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant randomized to Arm A (nivo+ipi) received the wrong treatment of chemo. This participant is counted in Arm A for baseline and efficacy analyses (analyses based on the randomized population) and is counted in Arm B (chemo) for exposure and safety analyses (based on the treated population). This participant was randomized prior to Revised Protocol 02 and is not included in the All Treated Participants from the Concurrently Randomized Arms B and C population.
Groups:
- Arm A: Nivo 3 mg/kg + Ipi 1 mg/kg: Participants received nivolumab 3 mg/kg IV over 30 minutes every 2 weeks for up to 3 doses (ie, 6 weeks of treatment; each cycle is 14 days). In Cycle 1 Day 1 only, nivolumab will be followed by a single dose of ipilimumab 1 mg/kg IV over 30 minutes.
  Following definitive surgery, participants could receive up to 4 cycles of adjuvant chemotherapy and/or radiation at the discretion of the investigator.
- Arm B: Platinum Doublet Chemo: Participants receive investigator-choice of platinum doublet chemotherapy regimens in 3-week cycles up to a maximum of 3 cycles of IV chemotherapy (ie, 9 weeks of treatment; each cycle is 21 days).
  Following definitive surgery, participants could receive up to 4 cycles of adjuvant chemotherapy and/or radiation at the discretion of the investigator.
- Arm C: Nivo 360 mg + Platinum Doublet Chemo: Participants receive nivolumab 360 mg IV + platinum doublet chemotherapy in 3-week cycles up to a maximum of 3 cycles of IV chemotherapy (ie, 9 weeks of treatment; each cycle is 21 days).
  Following definitive surgery, participants could receive up to 4 cycles of adjuvant chemotherapy and/or radiation at the discretion of the investigator.
Period: Randomization Period
Arm/Group | Arm A: Nivo 3 mg/kg + Ipi 1 mg/kg | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
Started | 113 | 213 | 179
All Concurrently Randomized Participants in Arms B and C (The primary population for efficacy analyses) | 0 | 179 | 179
Completed | 112 (One participant reassigned to Arm B as received the wrong treatment) | 207 | 176
Not Completed | 1 | 6 | 3
Not completed — Adverse event unrelated to study drug | 0 | 0 | 1
Not completed — Participant withdrew consent | 0 | 3 | 0
Not completed — Participant no longer meets study criteria | 1 | 3 | 2
Period: Neoadjuvant Treatment Period
Arm/Group | Arm A: Nivo 3 mg/kg + Ipi 1 mg/kg | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
Started | 111 | 208 | 176
All Treated Participants From Concurrently Randomized Arms B and C (The primary population for safety analyses) | 0 | 176 | 176
Completed | 101 | 177 | 165
Not Completed | 10 | 31 | 11
Not completed — Participant request to discontinue study treatment | 0 | 7 | 0
Not completed — Participant withdrew consent | 0 | 4 | 0
Not completed — Participant no longer meets study criteria | 0 | 1 | 0
Not completed — Disease progression | 3 | 2 | 1
Not completed — Study drug toxicity | 6 | 14 | 10
Not completed — Death | 1 | 0 | 0
Not completed — Adverse event unrelated to study treatment | 0 | 3 | 0
Period: Systemic Adjuvant Treatment Period
Arm/Group | Arm A: Nivo 3 mg/kg + Ipi 1 mg/kg | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
Started | 37 | 47 | 26
Completed | 28 | 41 | 22
Not Completed | 9 | 6 | 4
Not completed — Disease progression | 1 | 0 | 0
Not completed — Study drug toxicity | 4 | 5 | 1
Not completed — Adverse event unrelated to study drug | 1 | 0 | 1
Not completed — Participant request to discontinue treatment | 3 | 1 | 1
Not completed — Other reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivo 3 mg/kg + Ipi 1 mg/kg | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo | Total
Number analyzed (Participants) | 113 | 213 | 179 | 505
Age, Customized [Number; unit: Participants]
  < 65 | 62 | 99 | 93 | 254
  >= 65 AND < 75 | 40 | 96 | 75 | 211
  >= 75 AND < 85 | 11 | 17 | 11 | 39
  >= 85 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 65 | 51 | 156
  Male | 73 | 148 | 128 | 349
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 0 | 7
  Not Hispanic or Latino | 53 | 105 | 100 | 258
  Unknown or Not Reported | 58 | 103 | 79 | 240
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 41 | 96 | 86 | 223
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 4 | 13
  White | 64 | 108 | 89 | 261
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS)
Description: Event-free survival (EFS) is defined as the length of time from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on blinded independent central review (BICR) assessment per response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression, reoccurrence, or death due to any cause. (Up to a median of 30 months)
Population: All concurrently randomized participants in Arm C and Arm B
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
Number analyzed (Participants) | 179 | 179
Months | 20.80 [14.03 to 26.71] | 31.57 [30.16 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Arm B: Platinum Doublet Chemo vs Arm C: Nivo 360 mg + Platinum Doublet Chemo; Test type: Superiority; p = 0.0052, Log Rank; Stratified by PD-L1 (≥ 1% vs <1%/unevaluable/indeterminate), disease stage (IB/II vs IIIA), and sex (male vs female); Cox Proportional Hazard = 0.63, 97.38% CI 2-sided [0.43 to 0.91]

2. Primary Outcome: Pathologic Complete Response (pCR) Rate
Description: Pathologic complete response (pCR) rate is defined as the number of randomized participants with absence of residual tumor in lung and lymph nodes as evaluated by blinded independent pathological review (BIPR).
Time Frame: From randomization up to a median of 30 months after randomization.
Population: All concurrently randomized participants in Arm C and Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
Number analyzed (Participants) | 179 | 179
Participants | 4 | 43
Statistical Analysis 1: Comparison: Arm B: Platinum Doublet Chemo vs Arm C: Nivo 360 mg + Platinum Doublet Chemo; Test type: Superiority; % Difference = 21.6, 99% CI 2-sided [13.0 to 30.3] — Strata adjusted difference (Arm C - Concurrent Arm B) based on the CMH method of weighting. Stratified by PD-L1 (≥ 1% vs <1%/unevaluable/indeterminate), disease stage (IB/II vs IIIA), and sex (male vs female)
Statistical Analysis 2: Comparison: Arm B: Platinum Doublet Chemo vs Arm C: Nivo 360 mg + Platinum Doublet Chemo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 13.94, 99% CI 2-sided [3.49 to 55.75] — Strata adjusted odds ratio (Arm C over Concurrent Arm B) the Mantel-Haenszel method. Stratified by PD-L1 (≥ 1% vs <1%/unevaluable/indeterminate), disease stage (IB/II vs IIIA), and sex (male vs female)

3. Post Hoc Outcome: Event-Free Survival (EFS)
Description: as for outcome 1
Time Frame: From randomization to disease progression, reoccurrence, or death due to any cause. (Up to a median of 69 months)
Population: All concurrently randomized participants in Arm C and Arm B
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
Number analyzed (Participants) | 179 | 179
Months | 21.06 [16.53 to 36.76] | 59.60 [31.57 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Arm B: Platinum Doublet Chemo vs Arm C: Nivo 360 mg + Platinum Doublet Chemo; Test type: Superiority; Stratified by PD-L1 (≥ 1% vs <1%/unevaluable/indeterminate), disease stage (IB/II vs IIIA), and sex (male vs female); Cox Proportional Hazard = 0.68, 95% CI 2-sided [0.51 to 0.91]

4. Secondary Outcome: Major Pathologic Response (MPR) Rate
Description: Major pathologic response (MPR) rate is defined as number of randomized participants with </= 10% residual tumor in lung and lymph nodes as evaluated by blinded independent pathological review (BIPR). Viable tumors in situ carcinoma should not be included in MPR calculation.
Time Frame: From randomization up to a median of 30 months after randomization.
Population: All concurrently randomized participants in Arm C and Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
Number analyzed (Participants) | 179 | 179
Participants | 16 | 66
Statistical Analysis 1: Comparison: Arm B: Platinum Doublet Chemo vs Arm C: Nivo 360 mg + Platinum Doublet Chemo; Test type: Superiority; % Difference = 27.9, 95% CI 2-sided [19.6 to 36.1] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Arm B: Platinum Doublet Chemo vs Arm C: Nivo 360 mg + Platinum Doublet Chemo; Test type: Superiority; Odds Ratio (OR) = 5.70, 95% CI 2-sided [3.16 to 10.26] — Stratified by PD-L1 (≥ 1% vs <1%/unevaluable/indeterminate), disease stage (IB/II vs IIIA), and sex (male vs female)

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time between the date of randomization and the date of death. OS will be censored on the last date a participant was known to be alive.
Time Frame: From randomization to the date of death (Up to approximately 93 months)
Population: All concurrently randomized participants in Arm C and Arm B
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
Number analyzed (Participants) | 179 | 179
Months | 73.72 [47.34 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

6. Secondary Outcome: Time to Death or Distant Metastases (TTDM)
Description: TTDM is defined as the time between the date of randomization and the first date of distant metastasis or the date of death in the absence of distant metastasis. Distant metastasis is defined as any new lesion that is outside of the thorax using blinded independent central review (BICR) according to response evaluation criteria in solid tumors (RECIST) 1.1. Patients who have not developed distant metastasis or died at the time of analysis will be censored on the date of their last evaluable tumor assessment.
Time Frame: From randomization to the first date of distant metastasis or the date of death in the absence of distant metastasis (Up to approximately 84 months)
Population: All concurrently randomized participants in Arm C and Arm B
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
Number analyzed (Participants) | 179 | 179
Months | 36.76 [24.74 to 56.80] | 64.66 [49.02 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Arm B: Platinum Doublet Chemo vs Arm C: Nivo 360 mg + Platinum Doublet Chemo; Test type: Superiority; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.49 to 0.90] — Stratified by: PD-L1 status (≥ 1% vs <1%/not evaluable/indeterminate), disease stage (IB/II vs IIIA), and sex (male vs female)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from randomization to study completion (up to approximately 93 months). SAEs and Other AEs were assessed from first dose to 100days after the last dose of neoadjuvant therapy or 90 days after surgery, whichever is longer, and 30 days after the last dose of adjuvant therapy (up to approximately 5.5 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants (One participant randomized to Arm A (nivo+ipi) received the wrong treatment of chemo. This participant is counted in Arm B (chemo) safety analyses).
  The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Arm A: Nivo 3 mg/kg + Ipi 1 mg/kg | Arm B: Platinum Doublet Chemo | Arm C: Nivo 360 mg + Platinum Doublet Chemo
All-Cause Mortality (participants affected / at risk) | 46/112 | 105/214 | 66/179
Serious Adverse Events (participants affected / at risk) | 30/111 | 58/208 | 53/176
Other Adverse Events (participants affected / at risk) | 102/111 | 202/208 | 160/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivo 3 mg/kg + Ipi 1 mg/kg (N=111) | Arm B: Platinum Doublet Chemo (N=208) | Arm C: Nivo 360 mg + Platinum Doublet Chemo (N=176)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 6 | 3
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1
Ocular myasthenia (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Oesophageal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4
Death (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Pleural infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 5 | 8 | 6
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 1 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 2 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Immune-mediated myasthenia gravis (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 3
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic rupture (Vascular disorders) | 0 | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivo 3 mg/kg + Ipi 1 mg/kg (N=111) | Arm B: Platinum Doublet Chemo (N=208) | Arm C: Nivo 360 mg + Platinum Doublet Chemo (N=176)
Anaemia (Blood and lymphatic system disorders) | 9 | 78 | 62
Leukopenia (Blood and lymphatic system disorders) | 0 | 17 | 18
Neutropenia (Blood and lymphatic system disorders) | 1 | 39 | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 17 | 5
Atrial fibrillation (Cardiac disorders) | 0 | 8 | 9
Tinnitus (Ear and labyrinth disorders) | 1 | 17 | 6
Hyperthyroidism (Endocrine disorders) | 7 | 0 | 7
Hypothyroidism (Endocrine disorders) | 11 | 1 | 2
Constipation (Gastrointestinal disorders) | 24 | 73 | 63
Diarrhoea (Gastrointestinal disorders) | 18 | 34 | 21
Nausea (Gastrointestinal disorders) | 24 | 105 | 73
Stomatitis (Gastrointestinal disorders) | 4 | 12 | 6
Vomiting (Gastrointestinal disorders) | 10 | 30 | 20
Asthenia (General disorders) | 13 | 27 | 19
Fatigue (General disorders) | 24 | 39 | 30
Malaise (General disorders) | 3 | 26 | 27
Non-cardiac chest pain (General disorders) | 4 | 12 | 7
Oedema peripheral (General disorders) | 4 | 11 | 6
Pain (General disorders) | 8 | 29 | 18
Pyrexia (General disorders) | 18 | 23 | 20
Pneumonia (Infections and infestations) | 3 | 14 | 15
Upper respiratory tract infection (Infections and infestations) | 4 | 8 | 9
Incision site pain (Injury, poisoning and procedural complications) | 10 | 6 | 3
Procedural pain (Injury, poisoning and procedural complications) | 12 | 12 | 17
Wound complication (Injury, poisoning and procedural complications) | 4 | 15 | 14
Alanine aminotransferase increased (Investigations) | 7 | 18 | 13
Aspartate aminotransferase increased (Investigations) | 3 | 14 | 4
Blood creatinine increased (Investigations) | 1 | 14 | 15
Neutrophil count decreased (Investigations) | 7 | 46 | 28
Platelet count decreased (Investigations) | 2 | 14 | 18
Weight decreased (Investigations) | 3 | 12 | 10
White blood cell count decreased (Investigations) | 4 | 26 | 16
Decreased appetite (Metabolism and nutrition disorders) | 18 | 53 | 47
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 7 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 9 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 18 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 16 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 13 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 12 | 8
Dizziness (Nervous system disorders) | 10 | 10 | 9
Dysgeusia (Nervous system disorders) | 7 | 10 | 4
Headache (Nervous system disorders) | 8 | 16 | 8
Neuropathy peripheral (Nervous system disorders) | 0 | 4 | 10
Anxiety (Psychiatric disorders) | 8 | 8 | 4
Insomnia (Psychiatric disorders) | 8 | 15 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 31 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 18 | 15
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 30 | 18
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 28 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 7 | 13
Rash (Skin and subcutaneous tissue disorders) | 17 | 7 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02998528/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT02998528/SAP_001.pdf